CLINICAL TRIAL: NCT07374393
Title: Establishment of a Research Cohort on Sleep and Sleep Disorders in Patients With Neurological Diseases
Brief Title: Establishment of a Sleep and Sleep-disorder Research Cohort in Patients With Neurological Disorders
Status: Enrolling by invitation | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Zan Wang, Professor，Chief Physician, The First Hospital of Jilin University
Other Study IDs: SD-V01
Record Dates: First submitted 2026-01-14; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Sleep; Neurology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with neurological diseases: patients with confirmed diagnoses such as stroke, Parkinson's disease, epilepsy, cognitive disorders, neuroinfections, and immune-mediated neurological diseases
  Interventions: Other: Symptomatic and Etiological Treatment

INTERVENTIONS:
Other: Symptomatic and Etiological Treatment — sleep-related

SUMMARY:
This study aims to establish a research cohort on sleep and sleep disorders in patients with neurological diseases to systematically evaluate the relationship between various neurological conditions and sleep characteristics or disturbances.

DETAILED DESCRIPTION:
The cohort will include patients with confirmed diagnoses such as stroke, Parkinson's disease, epilepsy, cognitive disorders, neuroinfections, and immune-mediated neurological diseases, with collection of demographic data, medical history, and lifestyle factors. All participants will undergo standardized polysomnography (PSG), sleep questionnaires, assessments of cognition, mood, daytime function, as well as relevant imaging and laboratory tests. Designed as a prospective observational study, the cohort will focus on sleep architecture alterations, periodic limb movements, sleep-disordered breathing, REM sleep behavior disorder, nocturnal awakenings, heart rate, and oxygen saturation, and their associations with disease severity and progression. The data will provide a basis for exploring the mechanisms, early indicators, and potential interventions for sleep disturbances in neurological patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of neurological diseases, including but not limited to: Stroke (ischemic or hemorrhagic)，Parkinson's disease and other movement disorders，Epilepsy，Cognitive disorders (mild cognitive impairment or dementia)，Neuroinfections or immune-mediated neurological disorders
* Ability to complete standardized polysomnography, sleep questionnaires, and assessments of cognition, mood, and daytime function
* Voluntary participation and provision of written informed consent

Exclusion Criteria:

* Severe psychiatric disorders or unstable mental status precluding study assessments，Recent (within 3 months) serious infection, surgery, or major medical event
* Previously diagnosed severe primary sleep disorders (e.g., sleep apnea) under active treatment， -Pregnancy or lactation (if the study involves medication or interventions)

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Neurology patients able to undergo polysomnography examination
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-04 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Total sleep time measured by polysomnography | baseline, 3 months and one year
  Total sleep time is defined as the total amount of time spent asleep during the overnight polysomnography recording, expressed in minutes.
Wake after sleep onset measured by polysomnography | baseline, 3 months and one year
  Wake after sleep onset is defined as the total duration of wakefulness after sleep onset and before final awakening during the overnight polysomnography recording, expressed in minutes.
Sleep onset latency measured by polysomnography | baseline, 3 months and one year
  Sleep onset latency is defined as the time from lights off to the first epoch of sleep during overnight polysomnography.
Number of arousal events measured by polysomnography | baseline, 3 months and one year
  The number of arousal events is defined as the total number of arousals occurring during the overnight polysomnography recording.
Rapid eye movement sleep onset latency measured by polysomnography | baseline, 3 months and one year
  Rapid eye movement sleep onset latency is defined as the interval between sleep onset and the first occurrence of rapid eye movement sleep during the overnight polysomnography recording, expressed in minutes.
Non rapid eye movement sleep stage 1, 2, 3, and rapid eye movement sleep time measured by polysomnography | baseline, 3 months and one year
  Non-rapid eye movement (NREM) sleep stages 1, 2, and 3, and rapid eye movement (REM) sleep time are defined as the total duration spent in each sleep stage during overnight polysomnography, expressed in minutes.
Number of awakenings related to the event measured by polysomnography | baseline, 3 months and one year
  The number of awakenings related to respiratory events is defined as the total count of awakenings temporally associated with respiratory events during overnight polysomnography.
Number of respiratory events measured by polysomnography | baseline, 3 months and one year
  The number of respiratory events is defined as the total count of apnea and hypopnea events identified during overnight polysomnography.
Number of decreases in oxygen saturation measured by polysomnography | baseline, 3 months and one year
  The number of respiratory events is defined as the total count of respiratory events identified during overnight polysomnography.
Sleep period heart rate measured by polysomnography | baseline, 3 months and one year
  Sleep period heart rate is defined as the average heart rate measured during the sleep period as recorded by overnight polysomnography.
Number of rapid eye movement sleep without atonia measured by polysomnography | baseline, 3 months and one year
  The number of rapid eye movement sleep without atonia events is defined as the total count of rapid eye movement sleep epochs exhibiting increased muscle activity during overnight polysomnography.
Hypoxic burden measured by polysomnography | baseline, 3 months and one year
  Hypoxic burden is a quantitative measure of the cumulative severity of nocturnal hypoxemia, calculated from overnight polysomnography. It represents the total area under the curve of oxygen desaturation events, integrating both the depth and duration of oxygen desaturation across the entire sleep period.

SECONDARY OUTCOMES:
The score of Insomnia Severity Index scale | baseline, 3 months and one year
  The total score ranges from 0 to 28, and a higher score indicates higher levels of insomnia severity. A score of 8 or greater is the cut point for clinically possible insomnia.
The score of 14-item Hamilton anxiety rating scale | baseline, 3 months and one year
  The total score ranges from 0 to 56, and a higher score indicates higher levels of anxiety symptoms. A score of 7 or greater is the cut point for clinically possible anxiety.
The score of 17-item Hamilton depression rating scale | baseline, 3 months and one year
  The total score ranges from 0 to 52, and a higher score indicates higher levels of depression symptoms. A score of 7 or greater is the cut point for clinically possible depression symptom
The score of montreal cognitive assessment scale | baseline, 3 months and one year
  The total score ranges from 0 to 30, with higher scores indicating better global cognitive function. A score below 26 is commonly used as the cut-off for cognitive impairment.

OTHER OUTCOMES:
Plasma corticotropin-releasing factor level | baseline, 3 months and one year
  Plasma corticotropin-releasing factor concentration was measured as a biomarker of hypothalamic-pituitary adrenal axis activity. Higher levels indicate increased neuroendocrine stress response. Unit of Measure: pg/mL.
Plasma cortisol level | baseline, 3 months and one year
  Plasma cortisol concentration was assessed as an indicator of hypothalamic-pituitary-adrenal axis function. Higher levels reflect increased physiological stress response. Unit of Measure: μg/dL.
Serum interleukin-6 level | baseline, 3 months and one year
  Serum interleukin-6 concentration was measured as a marker of systemic inflammation. Higher levels indicate greater inflammatory activity. Unit of Measure: pg/mL.
Serum brain-derived neurotrophic factor level | baseline, 3 months and one year
  Serum brain-derived neurotrophic factor concentration was measured as a biomarker associated with neuroplasticity and neuronal function. Higher levels indicate enhanced neurotrophic activity. Unit of Measure: pg/mL.
Gray matter volume measured by structural magnetic resonance Imaging | baseline, 3 months and one year
  Gray matter volume was derived from T1-weighted structural MRI using voxel-based morphometry, reflecting regional brain tissue volume.
Cortical thickness measured by structural magnetic resonance Imaging | baseline, 3 months and one year
  Cortical thickness was quantified from T1-weighted MRI as the distance between the white matter and pial surfaces, reflecting cortical integrity.
Hippocampal volume measured by structural magnetic resonance Imaging | baseline, 3 months and one year
  Hippocampal volume was extracted from T1-weighted MRI using automated segmentation and normalized for intracranial volume.
Resting-state functional connectivity measured by resting-state functional magnetic resonance imaging | baseline, 3 months and one year
  Functional connectivity was assessed by calculating temporal correlations of blood-oxygen-level-dependent signals between predefined brain regions during rest.
Amplitude of low-frequency fluctuation measured by resting-state functional magnetic resonance | baseline, 3 months and one year
  Amplitude of low-frequency fluctuation reflects the amplitude of spontaneous low-frequency BOLD signal oscillations, indicating regional intrinsic neural activity.
Regional homogeneity measured by resting-state functional magnetic resonance | baseline, 3 months and one year
  Regional homogeneity was calculated to assess the similarity of the time series of a given voxel with its neighboring voxels, reflecting local synchronization of brain activity.
Global blood-oxygen-level-dependent signal measured by resting-state functional magnetic resonance | baseline, 3 months and one year
  The global blood-oxygen-level-dependent signal represents the average blood-oxygen-level-dependent signal across the whole brain, reflecting the overall amplitude and synchronization of brain activity.
Fractional anisotropy measured by diffusion tensor imaging | baseline, 3 months and one year
  Fractional anisotropy reflects the degree of directional water diffusion and was used to assess white matter microstructural integrity.
Mean diffusivity measured by diffusion tensor imaging | baseline, 3 months and one year
  Mean diffusivity quantifies the overall magnitude of water diffusion and reflects microstructural tissue changes.
Cerebrospinal fluid flow dynamics measured by resting-state functional magnetic resonance | baseline, 3 months and one year
  Cerebrospinal fluid flow dynamics were assessed using MRI-based methods to characterize CSF motion and pulsatility.
Phase difference of dynamic cerebral autoregulation | baseline, 3 months and one year
  Dynamic cerebral autoregulation was assessed using the phase difference between cerebral blood flow velocity and arterial blood pressure fluctuations. Larger phase differences indicate better autoregulatory function.
Gain of dynamic cerebral autoregulation | baseline, 3 months and one year
  Gain represents the magnitude of cerebral blood flow velocity changes in response to blood pressure fluctuations, with lower gain values indicating more effective autoregulation.

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No